CLINICAL TRIAL: NCT03182140
Title: KYleena Satisfaction Study / Observational Study on User Satisfaction With the Levonorgestrel Intrauterine Delivery System Kyleena (LNG-IUS 12) in New Contraceptive Users and After Switching From Another Contraceptive Method
Acronym: KYSS
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19186
Record Dates: First submitted 2017-05-19; First posted 2017-06-09 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Contraception
Keywords: long-acting contraception,; unintended pregnancy; satisfaction; bleeding profile; amenorrhea
MeSH Terms: conditions — Personal Satisfaction; Amenorrhea | interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kyleena: Non-interventional, observational, uncontrolled study in women that have chosen Kyleena as their contraceptive method before entering the study
  Interventions: Drug: Kyleena

INTERVENTIONS:
Drug: Kyleena — Kyleena - intrauterine delivery system containing 19.5 mg LNG

SUMMARY:
The main goal of this non-interventional study (NIS) is to evaluate user satisfaction with Kyleena in a real-life setting and to identify factors which influence user satisfaction, taking into account previously used contraceptive methods and reasons for use of Kyleena.

ELIGIBILITY:
Inclusion Criteria:

* Women requesting contraception with Kyleena. The woman's informed decision for contraception with Kyleena was made before and independently from the study as per investigator's routine practice
* Written informed consent.

Exclusion Criteria:

* Contraindications for Kyleena according to the local market authorization/SmPC
* Mental incapacity to consent and provide data during the observational study
* Women participating in an investigational program with interventions outside of routine clinical practice.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women in the respective participating country requesting contraception with Kyleena will be eligible to be enrolled.
  Women can be screened for the study only after an informed decision for Kyleena has been made by the woman and the treating health care professional such as her physician/gynecologist or midwife. Indication and contraindications according to the local market authorization/ summary of product characteristics (SmPC) should be carefully considered.
Sampling Method: Non-Probability Sample
Enrollment: 1134 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction with Kyleena assessed by questionnaire | approximately at 12 months after insertion or at premature discontinuation
  The rating is based on the 5-item Likert scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied).

SECONDARY OUTCOMES:
Overall satisfaction with Kyleena assessed by questionnaire | approximately 4-12 weeks after insertion
  The rating is based on the 5-item Likert scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied).
Ease of insertion assessed by investigator | Day 1
  The rating is based on the categories easy, slightly difficult, very difficult.
Pain at insertion assessed by participant | Day 1
  The rating is based on the categories none, mild, moderate, or severe
Satisfaction with the menstrual bleeding profile with Kyleena assessed by questionnaire | after approximately 12 months or at premature discontinuation and approximately 4-12 weeks after insertion
  Satisfaction with the menstrual bleeding profile with Kyleena assessed by women who did and did not experience menstrual bleeding during the last three months when answering the question "How satisfied were you with your menstrual bleeding pattern?" respectively.
  The rating is based on the 5-item Likert scale (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied).

CONTACTS AND LOCATIONS:
Locations (19):
- United States (12):
  - Jennifer Grube, MD, FACOG, Lakewood, Colorado
  - Physician Care Clinical Research LLC, Sarasota, Florida
  - Visions Clinical Research, Wellington, Florida
  - New England Center for Clinical Research Primacare Research, LLC, Fall River, Massachusetts
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Lawrence OB/GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - ProHEALTH Care Associates, Port Jefferson, New York
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Radiant Research, Akron, Ohio
  - TMC Life Research, Houston, Texas
  - Physician's Research, Draper, Utah
  - Physician's Research Options LLC - Revere Women's Health OB/GYN Clinic, Pleasant Grove, Utah
- Many locations, Multiple Locations, Belgium
- Many locations, Multiple Locations, Canada
- Many locations, Multiple Locations, Germany
- Many locations, Multiple Locations, Mexico
- Many locations, Multiple Locations, Norway
- Many locations, Multiple Locations, Spain
- Many locations, Multiple Locations, Sweden

REFERENCES:
- [Derived] Romer T, Frenz AK, Dietrich-Ott S, Fiedler A. The use of LNG-IUS-19.5 mg in daily gynecological routine practice in Germany: data from the Kyleena Satisfaction Study (KYSS). Arch Gynecol Obstet. 2024 May;309(5):2021-2030. doi: 10.1007/s00404-024-07421-5. Epub 2024 Feb 29. PMID 38421421
- [Derived] Stovall DW, Aqua K, Romer T, Donders G, Sordal T, Hauck B, Llata ES, Kallner HK, Salomon J, Zvolanek M, Frenz AK, Bohnke T, Bauerfeind A. Satisfaction and continuation with LNG-IUS 12: findings from the real-world kyleena(R) satisfaction study. Eur J Contracept Reprod Health Care. 2021 Dec;26(6):462-472. doi: 10.1080/13625187.2021.1975268. Epub 2021 Sep 16. PMID 34528857
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/